CLINICAL TRIAL: NCT00722163
Title: A Randomized Controlled Trial of Individual Therapy for First Episode Psychosis
Acronym: PSTEP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ontario Mental Health Foundation (Other Government)
Collaborators: Schizophrenia Society of Ontario (Other)
Responsible Party: Dr. Jean Addington, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 195/2006; NCT00495911 (obsolete NCT alias)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Psychosis
Keywords: Cognitive Behavioural therapy; Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): behavioural
  Interventions: Other: Cognitive Behavioural Therapy
- 2 (Active Comparator): befriending
  Interventions: Other: befriending
- 3 (No Intervention): TAU

INTERVENTIONS:
Other: Cognitive Behavioural Therapy
  Arms: 1
Other: befriending
  Arms: 2

SUMMARY:
In the first year of treatment after a FE of SCZ, 75% to 90% of patients achieve remission from psychotic symptoms. However, approximately 40% of FE patients are non-adherent to medication regimes and more than 60% have intermittent periods of gaps of non-adherence. Relapse rates are high with 82% of patients relapsing at least once within 5 years. Unfortunately even amongst those who do achieve full remission from psychotic symptoms, functional recovery remains a major challenge for patients. All the evidence suggests that individuals with SCZ do best with a combination of pharmacology and psychosocial intervention. Cognitive-behavior therapy (CBT) is gaining recognition as an effective treatment in SCZ and is in fact the only psychosocial treatment in SCZ with proven durability at short term follow-up. Although it is currently being used, the investigators need to learn more about the impact of CBT on FE SCZ especially as experts are advocating for CBT to be a critical component of FE clinical services.

DETAILED DESCRIPTION:
The primary problem to be addressed is the incomplete functional recovery following a FE of SCZ and whether CBT is an effective treatment to aid this recovery. If CBT were to positively impact recovery in the FE we then need to address (i) which mechanisms are responsible for this improvement, and (ii) whether this treatment is effective for all FE patients.

ELIGIBILITY:
Inclusion Criteria:

1. stabilized outpatients,
2. ages 16 to 35
3. meet DSM-IV criteria for: schizophrenia, schizophreniform disorder, brief psychotic disorder, delusional disorder, schizoaffective disorder, substance induced psychotic disorder, or psychotic disorder NOS. Participants who also meet DSM-IV criteria for substance abuse or dependence will not be excluded.
4. are competent and willing to give consent
5. are within 12 months of admission to the FEPP for a FE.

Exclusion:

1. serious risk of suicide or violence to others
2. a primary diagnosis of drug-induced psychosis or psychosis due to a general medical condition.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-05 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Social Functioning | 18 months
Positive & negative symptoms | 18 months
Individual dimensions of psychotic symptoms | 18 months
Depression | 18 months
Substance use | 18 months
Alcohol and Drug Use | 18 months
Medication adherenceAdaptation to illness | 18 months
Self Esteem | 18 months
Coping Skills (MACS) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Addington, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada